CLINICAL TRIAL: NCT01763775
Title: Verify the Functions and Efficiency of Transtek (Trade Mark) Body Fat Analyzer, GBF-1251-B, BF-1255-B, BF-1256-B, and GBF-1257-B
Brief Title: Clinical Trial of Transtek Body Fat Analyzer (GBF-1251-B & Other 3 Models)
Acronym: BS-BT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leo Wang (Other)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor-Investigator, Leo Wang, Team Leader, BTS International
Organization: BTS International (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None
Other Study IDs: 13001_Body Scale; BTS13001 (Other: BTSInternational)
Record Dates: First submitted 2013-01-05; First posted 2013-01-09 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2013-01

CONDITIONS: Weight; Body Fat Disorder; Bone Mass
Keywords: weight; total body water; body fat; muscle mass; bone mass
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transtek 125X (Experimental): Which measured by DUT (Transtek 125X): GBF-1251-B, BF-1255-B, BF-1256-B, GBF-1257-B.
  Interventions: Device: Transtek 125X; Device: Transtek 950D
- Transtek 950D (Experimental): Measured by Reference (Transtek 950D): GBF-950-D.
  Interventions: Device: Transtek 125X; Device: Transtek 950D

INTERVENTIONS:
Device: Transtek 125X — Measuring weight, total body water, body fat, muscle mass, and bone mass. Measure each participants by Transtek 125X (GBF-1251-B, BF-1255-B, BF-1256-B, GBF-1257-B).
Device: Transtek 950D — Measuring weight, total body water, body fat, muscle mass, and bone mass. Measure each participants by Transtek 950D (GBF-950-D).

SUMMARY:
The clinical protocol of the clinical testing of this device:

1. Objective of the test: To verify the functions and efficiency of devices.
2. Test methods and procedures: Comparison Test.
3. Device Under Test (DUT): Transtek Body Fat Analyzer, Model: GBF-1251-B, BF-1255-B, BF-1256-B, and GBF-1257-B.
4. Comparison device: Transtek, Glass Body Fat Analyzer, GBF-950-D.
5. Study endpoints: DUT and the comparison device are substantial equivalence.
6. Statistical methodology used: Description of statistical methods.

DETAILED DESCRIPTION:
1. Test Purpose:

   The aim of clinical test is to collect weight, body fat, total body water, bone mass, and muscle mass reading value which measured by DUT and reference device.
2. Target Subject:

   The subject database shall contain at least 25 male and 25 female subjects and all above 18 years old.
3. Test procedures:

   1. Record the name, age, gender, and height of each subject.
   2. Let subject seated calmly for two minutes before test, dry the feet.
   3. Use device to measure weight, body fat, total body water, bone mass, and muscle mass; record reading value.
   4. For each subject, repeat 3) to get 3 pairs measurements.
   5. Repeat step 1) to 4) for every device (DUT: GBF-1251-B, BF-1255-B, BF-1256-B, and GBF-1257-B; and reference device: GBF-950-D).
   6. Repeat step 1) to 5) for each subject.
4. Note:

   1. No motion and speaking are allowed during the measurement.
   2. All DUT use the same algorithms and contact the patient at the same body locations (feet), and operate on the same frequency.
   3. Test environment: Temperature: 22±1℃; Relative humidity: 40~70%.

ELIGIBILITY:
Inclusion Criteria:

* male,female

Exclusion Criteria:

* below 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
BMI (Body Mass Index) | 5 Day
  Body Fat, Total Body Water, Muscle Mass, Bone Mass

SECONDARY OUTCOMES:
Weight | 5 Days
  Body Weight

CONTACTS AND LOCATIONS:
Overall Officials: Guoqing Li, Director, Principal Investigator — Wuhou District Hospital
Locations (1):
- Wuhou District Hospital, Chengdu, Sichuan, China